CLINICAL TRIAL: NCT05584241
Title: Behavioral Change Following Culturally Informed Biomarker Disclosure in Alzheimer's Disease
Brief Title: Behavioral Change Following Alzheimer's Disease (AD) Biomarker Disclosure
Acronym: SHARED III
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Annalise Rahman-Filipiak, Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00221221; 1K23AG070044-01 (NIH)
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Amnestic Mild Cognitive Disorder
Keywords: AD Biomarkers; Alzheimer's Disease; Mild Cognitive Impairment; Amnestic Mild Cognitive Disorder
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Randomized delayed start design. Participants are randomized to receive, at baseline, either 'Diagnostic Disclosure Protocol' (cognitive testing/diagnosis) with an option to receive biomarker results after 6 months or 'Biomarker Disclosure Protocol' (cognitive testing, diagnosis, positron emission tomography-based amyloid and tau imaging. They are further categorized by biomarker status (+/positive or -/negative) for reporting purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diagnostic Disclosure (Active Comparator): Personalized disclosure on cognitive test results and research diagnosis, plus post-disclosure dementia risk reduction counseling.
  For reporting purposes those participants randomized to this condition are analyzed by biomarker status (positive/+ or negative/-).
  Interventions: Behavioral: Diagnostic Disclosure Protocol
- Biomarker and Diagnostic Disclosure (Experimental): Participants receive information about their cognitive test results and research diagnosis. In addition, participants receive information about whether they currently have elevated or not-elevated amyloid and/or tau based on recent PET imaging. PET is a type of imaging biomarker (Aß-PET and tau PET) for clinical diagnosis of Alzheimer's disease. These actions are followed by post-disclosure dementia risk reduction counseling.
  For reporting purposes those participants randomized to this condition are analyzed by biomarker status (positive/+ or negative/-).
  Interventions: Behavioral: Biomarker Disclosure Protocol

INTERVENTIONS:
Behavioral: Diagnostic Disclosure Protocol — Personalized disclosure on cognitive test results and research diagnosis, plus post-disclosure dementia risk reduction counseling.
  Arms: Diagnostic Disclosure
Behavioral: Biomarker Disclosure Protocol — Participants receive information about their cognitive test results and research diagnosis just like in the diagnostic disclosure protocol. In addition, participants receive information about whether they currently have elevated or not-elevated amyloid and/or tau based on recent PET imaging. PET is a type of imaging biomarker (Aß-PET and tau PET) for clinical diagnosis of Alzheimer's disease. These actions are followed by post-disclosure dementia risk reduction counseling.
  Arms: Biomarker and Diagnostic Disclosure

SUMMARY:
The proposed project will assess long-term changes to health/lifestyle, advanced planning, and research engagement that Black and White patients with Amnestic Mild Cognitive Impairment (aMCI) make following disclosure of positron emission tomography-based amyloid and tau burden and associated risk of conversion to Dementia-Alzheimer's Type. Healthcare access will be explored as potential barrier to or facilitator of behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Amnestic Mild Cognitive Impairment within the past 12 months,
* Available PET Aβ and tau imaging

Exclusion Criteria:

* Significant neurologic diagnosis (e.g., Alzheimer's dementia or other neurodegenerative dementia, Parkinson's disease, seizure disorder, tumor, multiple sclerosis)
* Neurologic injury (e.g., significant stroke or moderate-severe head injury, defined by loss of consciousness > 5 minutes, presence of significant post-traumatic amnesia, or the need for extended hospitalization or intervention)
* Motor abnormalities indicative of a non-AD etiology
* Severe mental illness (e.g., bipolar disorder, psychosis), moderate-severe mood or anxiety disorder, active substance use disorder (o reduce the likelihood of severe psychological distress, participants must screen negative for moderate-severe depressive or anxiety symptoms at study enrollment.)
* Inability to provide independent informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Post-disclosure health behavior change as measured by the health behavior subscale score | 6 months
  Subscale is a part of the Stages of Change Interview. Respondents will rate seven items relating to behavioral changes they have made post-disclosure on a Likert scale ranging from 1 = "I have not considered/am not interested in making this change" to 5 = "I have already made and maintained this change." Subscale score total ranges from 7 to 35 with higher scores indicating more engagement.
Post-disclosure health behavior change as measured by the health communication subscale score | 6 months
  Subscale is a part of the Stages of Change Interview. Respondents will rate two items relating to health communication using a Likert scale. Subscale score total ranges from 2 to 10 with higher scores indicating more engagement.
Post-disclosure health behavior change as measured by the advanced planning subscale score | 6 months
  Subscale is a part of the Stages of Change Interview. Respondents will rate seven items relating to advanced planning using a Likert Scale. Subscale score total ranges from 7 to 35 with higher scores indicating more engagement.
Post-disclosure health behavior change as measured by the research engagement subscale score | 6 months
  Subscale is a part of the Stages of Change Interview. Respondents will rate one item relating to research engagement on a Likert scale. Subscale score total ranges from 1 to 5 with higher scores indicating more engagement.
Percent participant retention in University of Michigan Memory and Aging Project (UMMAP) study | Up to 24 months
  Measured by attendance at study visits

CONTACTS AND LOCATIONS:
Overall Officials: Annalise Rahman-Filipiak, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No